CLINICAL TRIAL: NCT02289235
Title: The Effects of Ginger on Biochemical Markers and Imaging Studies of Patients With Type 2 Diabetes Mellitus and Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Effects of Ginger on Nonalcoholic Fatty Liver Disease in T2DM
Acronym: GinLivDM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal Medicine & Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P-9364-6254
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Fatty Liver; Diabetes Mellitus, Type 2
Keywords: Ginger; Medicine, traditional; Herbal medicine
MeSH Terms: conditions — Fatty Liver; Diabetes Mellitus, Type 2 | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger (Experimental): Ginger powder capsule 500 mg
  Interventions: Drug: Ginger
- Placebo (Placebo Comparator): Placebo powder capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger — Ginger powder capsule 1000 mg twice daily for 3 months
  Arms: Ginger
Drug: Placebo — Placebo powder 2 capsules twice daily for 3 months
  Arms: Placebo

SUMMARY:
The investigators want to evaluate the effects and safety of ginger in treatment of nonalcoholic fatty liver disease (NAFLD) in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Ginger (Zingiber officinale Roscoe) has been cultivated for medicinal and culinary purposes for at least two millennia. It contains several hundred valuable compounds and new constituents are still being found. Ginger's high antioxidant value has proved highly effective with its ability to scavenge a number of free radicals and protect cell membrane lipids from oxidation in a dose-dependent manner.

In a randomized double-blind placebo-controlled clinical trial, the investigators want to investigate the effects of ginger in treatment of nonalcoholic fatty liver disease (NAFLD) in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Controlled type 2 diabetes mellitus (HbA1c<7%)
* Age: 20-65 years
* Body mass index: 18-35 kg/m2
* Serum ALT level: >60 U/Lit. in males, >38 U/Lit. in females
* Grade >=2 fatty liver in liver sonography

Exclusion Criteria:

* Pregnancy
* Acute or chronic liver failure
* Acute or chronic renal failure
* Autoimmune or viral hepatitis
* Wilson's disease
* Alcoholism
* Malignancy
* Hypothyroidism or hyperthyroidism
* Drug used in last three months: OCP, vitamin E, ursodeoxycholic acid, glucocorticoids.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in ALT (liver transaminases) level | Baseline and 3 months
  Change in the concentration of ALT (liver transaminases)
Change in score of fatty liver in fibroscan | Baseline and 3 months
  Change in score of fatty liver in fibroscan (elastography)

SECONDARY OUTCOMES:
Change in AST (liver transaminases) level | Baseline and 3 months
  Change in the concentration of AST (liver transaminases)
Change in Gama GT (γ-glutamyl transpeptidase) levels | Baseline and 3 months
  Change in the concentration of Gama GT (γ-glutamyl transpeptidase)
Number of patients with adverse events | 4 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mesbah Shams, M.D., Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Majid Nimruzi, M.D., Principal Investigator — Research Center for Traditional Medicine, Shiraz University of Medical Sciences; Kamran Bagheri Lankarani, M.D., Principal Investigator — Health policy Research Center, Shiraz University of Medical Sciences; Parisa-sadaat Ghoreishi, M.D., Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No